CLINICAL TRIAL: NCT04025983
Title: Effectiveness of GastimunHp Plus in Supporting the Treatment of Peptic Ulcer Disease With Helicobacter Pylori Infection
Acronym: GasHp
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was slow and disrupted by COVID-19.
Sponsor: Institute of Gastroenterology and Hepatology, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TH1903
Record Dates: First submitted 2019-07-12; First posted 2019-07-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Helicobacter Pylori Infection; Peptic Ulcer
Keywords: Helicobacter pylori; peptic ulcer; Lactobacillus johnsonii; immunoglobin Y
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational product (IP) is compared with a placebo. The IP and placebo are manufactured by the sponsor and then sent to the trial pharmacist. They are only different in a number in the package label, and only the sponsor knows which number is the IP and will call them "product I" and "product II". This labelling is not revealed to the study team, the trial pharmacist, and the biostatistician.
  In the random number sequences generated by the biostatistician, the study numbers will be allocated to either "product I" or "product II". The trial pharmacist is responsible for making product bags using study numbers and allocation given by the biostatistician. The product bags are transferred to the study team. In this way, the study team and patients are completely masked to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GastimunHp Plus (Experimental): 1 sachet of GastimunHp Plus twice daily during or after meals.
  Interventions: Dietary Supplement: GastimunHp Plus
- Placebo (Placebo Comparator): 1 sachet of placebo twice daily during or after meals.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: GastimunHp Plus — Each sachet contains 6mg of IgY and 50 mg of heat-killed Lactobacillus johnsonii No. 1088.
  Arms: GastimunHp Plus
Other: Placebo — The placebo contains neither IgY nor L. johnsonii.
  Arms: Placebo

SUMMARY:
Challenges in the treatment of Helicobacter pylori (H. pylori) include increasing antimicrobial resistance and patient's low tolerance to some regimens. Lactobacillus johnsonii (L. johnsonii) and Immunoglobulin Y (IgY) have been shown to decrease the amount and activity of H. pylori in human stomach and can increase patient's tolerance. We conduct a single-center double-masked randomized controlled trial to evaluate the effectiveness of GastimunHp Plus (a product combining L. johnsonii and IgY) in improving the clearance of H. pylori after six to eight weeks of treatment and side effects of H. pylori treatment. H. pylori is tested by C13- or C14-urea breath test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gastritis, duodenitis, or peptic ulcer.
* Tested positive with Helicobacter pylori using C13- or C14-urea breath test or urease test.
* Indicated for Helicobacter pylori eradication.

Exclusion Criteria:

* Suspected malignant lesions.
* Children under 10 years of age; pregnant or lactating women.
* Allergic to chicken egg.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with negative urea breath test after 6-8 weeks | Six to eight weeks after recruitment
  Patients tested negative with Helicobacter pylori using C13- or C14-urea breath test.

SECONDARY OUTCOMES:
Proportion of patients with clinical improvement after 6-8 weeks | Six to eight weeks after recruitment
  Symptom resolution evaluated clinically.
Proportion of patients with adverse effects | Six to eight weeks after recruitment
  Any adverse effects that are deemed related to the investigational product.
Proportion of patients with improvement of lesions on endoscopy | Six to eight weeks after recruitment
  Improvement of lesions detected on baseline on upper gastrointestinal endoscopy. Improvement was determined by expert's opinion.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Gastroenterology and Hepatology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided